CLINICAL TRIAL: NCT03396055
Title: Investigation of the Relationship Between Surgical Approaches, Psychological Intervention, Neuromuscular Control, Rehabilitation Exercise and Biomechanical Characteristics in Radiculomyelopathy Patients
Brief Title: Investigation in Integrated Perspective of Radiculomyelopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201505093RINA
Record Dates: First submitted 2017-12-26; First posted 2018-01-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-04

CONDITIONS: Cervical Myelopathy; Cervical Radiculopathy
Keywords: decompression surgery; functional outcome; biomechanic; rehabilitation
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Specific rehabilitation exercise
  Interventions: Other: specific rehabilitation exercise
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: specific rehabilitation exercise — specific rehabilitation exercise for patients with cervical myelopathy
  Arms: Treatment group

SUMMARY:
Cervical radiculopathy and myelopathy are common degenerative disorders, which can create a large amount of social and medical burden. The aims of this study are(1) to investigate the functional outcomes progression before and after surgery, (2) to evaluate the biomechanical change and compensatory patterns of patients with or without decompression surgery, and (3) to design innovation intervention for the patients with cervical myelopathy and radiculopathy.

DETAILED DESCRIPTION:
Neck pain, which is common in population recently, is causing the huge burden in the global medical service system. Cervical myelopathy, that is induced by disc degeneration, is turning to be an alarming public health issue. The clinical manifestations of cervical myelopathy include neck/shoulder pain, numbness/weakness of four limbs, sensorimotor impairment, and sociopsychological dysfunction. However, most of the previous studies tend to justify patients, prognosis in a single dimension. The investigators realized that no standard protocol for management in patients with the variety of manifestation and severity of signs and symptoms.This study is purposed to integrate and analyze the finding in surgery selection, clinical manifestation, psychological consultation, compensatory patterns in the neuromusculoskeletal system, postural control, home exercise and biomechanical features. Then, the investigators will develop a complementary model in assessment and prediction of prognosis, and also an applicable standard guideline in the clinical setting. To achieve the expected target, the principal investigator will play the role as the main coordinator in the team. The 3-year plan is listed as below:

1. In the first year, the patients will be recruited for projects from different co-investigators. The recruited participants will be allocated to different study group after assessment to ensure the most suitable intervention are offered to the participants.
2. In the second year, the participants' recruitment will be continuing. The effectiveness previous treatment will be assessed. The study procedure will be adjusted based on pilot results.

2. In the third year, the study finding of all co-investigators and results of the biomechanical analysis will be integrated to establish the model of prognosis prediction and clinical management guideline. This study will provide a complete clinical management guideline in cervical myelopathy, which is expected to be globally leading reference in the management of cervical myelopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as cervical myelopathy or radiculopathy based on imaging results

Exclusion Criteria:

* With spondylolisthesis, rheumatoid arthritis, multiple sclerosis
* With cancer/tumor
* With neurological or psychological disorder
* Not suitable for cervical decompression surgery or physical therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 1 year
  Questionnaire
Japanese Orthopaedic Association Myelopathy Evaluation Questionnaire (JOACMEQ) | 1 year
  Questionnaire
Modified Japanese Orthopaedic Association Scale (Modified JOA scale) | 1 year
  Investigator-administered scale Sub-scale 1: Motor Dysfunction score of the upper extremity (maximum score-5, minimum score-0) Sub-scale 2: Motor Dysfunction score of the lower extremity (maximum score-7, minimum score-0) Sub-scale 3: Sensory dysfunction score of the upper extremities (maximum score-3, minimum score-0) Sub-scale 4: Sphincter dysfunction (maximum score-3, minimum score-0) Higher score shows better outcome
Nurick scale | 1 year
  Investigator-administered scale The total maximum score is 5: the total minimum score is 0. Higher score shows worse outcome
Grip and release test | 1 year
  Functional movement
Foot taping test | 1 year
  Functional movement
5 times sit to stand | 1 year
  Functional movement
10 second step test | 1 year
  Functional movement
Kinetic variables | 1 year
  The ground reaction force, moment and center of pressure recorded by force platform during standing and ambulation.
Neuropathic Pain Symptom Inventory | 1 year
  Questionaire
Magnetic Resonance Imaging (MRI) | 1 year
  The cortical network of patients assessed by Diffusion Spectrum Imaging of the brain
SF-36 | 1 year
  Questionnaire
WHOQOL_BREF | 1 year
  Questionnaire
Kinematic variables | 1 year
  Range of motion
Muscle activities in Electromyography (EMG) | I year
  Muscle activities in neck and lower limbs

CONTACTS AND LOCATIONS:
Overall Officials: Dar-Ming Lai, Ph.D, Principal Investigator — National Taiwan Unversity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin IS, Lai DM, Ding JJ, Chien A, Cheng CH, Wang SF, Wang JL, Kuo CL, Hsu WL. Reweighting of the sensory inputs for postural control in patients with cervical spondylotic myelopathy after surgery. J Neuroeng Rehabil. 2019 Jul 25;16(1):96. doi: 10.1186/s12984-019-0564-2. PMID 31345240